CLINICAL TRIAL: NCT02172183
Title: Group Therapy for Adolescents With Attention-Deficit/Hyperactivity Disorder: a Randomized Multicenter Controlled Trial
Brief Title: CBT Group for Adolescents With ADHD: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Principal Investigator, Raquel Vidal, PhD, Hospital Universitari Vall d'Hebron Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT-RV
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: cognitive-behavioral therapy, adolescents, ADHD.
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT group (Experimental): This group consist on a combined intervention: CBT group + psychopharmacological treatment. The group program was based on cognitive-behavioral principles and also motivational interviewing techniques to facilitate skills implementation. The treatment comprised 12 manualized sessions with an inattention module and an impulsivity module.
  Interventions: Behavioral: CBT group
- Psychopharmacological treatment (Active Comparator): Participants were only visited to monitor their adherence and continuation on medications for ADHD (methylphenidate or atomoxetine) as prescribed by their psychiatrist.
  Interventions: Drug: Psychopharmacological treatment

INTERVENTIONS:
Drug: Psychopharmacological treatment — methylphenidate or atomoxetine
  Arms: Psychopharmacological treatment
Behavioral: CBT group
  Arms: CBT group

SUMMARY:
This is the first randomized controlled study that tests the efficacy of a cognitive-behavioral group therapy (CBT) on adolescents with ADHD who were in pharmacological treatment but still presented persistent symptoms.

DETAILED DESCRIPTION:
A multicenter, randomized rater-blinded controlled trial was carried out in a sample of 119 adolescents (15-21 years) and was conducted between April 2012- May 2014. Patients were randomly assigned to 12 group manualized cognitive-behavioural group therapy sessions (n=45) or a waiting list control group (N=44). Primary outcomes were assessed by a blind evaluator (ADHD Rating Scale, Clinical Global Impression Scale for Severity, Global Assessment Functioning) before and after treatment as well as by self-report and parent informant ratings.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV ADHD diagnosis
* age between 15 and 21 years
* stabilized doses of medication for ADHD for at least 2 months prior to the study
* agreement not to seek out any other psychiatric or psychological treatment during the study.

Exclusion Criteria:

* affective disorders
* anxiety disorders
* psychotic disorders
* personality disorders
* substance use disorders in the past 6 months
* pervasive developmental disorder
* patients with an IQ lower than 85
* patients receiving concurrent psychological interventions.

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Post-treatment ADHD symptoms | Post-treatment (after receiving 3 month treatment)
  measured by ADHD Rating Scale (clinician-administered version for the adolescent and also parent informant). It is a 18 item scale which assesses the diagnostic criteria for ADHD and rates the frequency of each item on a 4 point Likert scale.
Post-treatment functional impairment | Post-treatment (after receiving 3 month treatment)
  Assessed by Weiss Functional Impairment Scale (WFIRS) self report and parent version (an appropriate measure for functional impairment associated with ADHD) and by GAF (Global Assessment of Functioning) evaluated by a blinded rater. It is a clinician-administered measure to assess clinical severity and functioning.

SECONDARY OUTCOMES:
Post-treatment depression symptoms | Post-treatment (after receiving 3 month treatment)
  assessed by Beck Inventory Depression Scale (BDI). It is a 21 item scale to test depression symptoms where respondents rate how they have been feeling during the past week on a 4 point Likert scale (0-3)
Post-treatment anxiety symptoms | Post-treatment (after receiving 3 month treatment)
  assessed by State-Trait Anxiety Inventory. It is a 40 item scale. It differentiates between the temporary condition of "state anxiety" and the more general and long-standing quality of "trait anxiety".
Post-treatment anger management | Post-treatment (after receiving 3 month treatment)
  State-Trait Anger Expression Inventory-2 (STAXI-2)was used for patients between 16-21 years and STAXI-NA for 15 years-old patients. The STAXI-2 is a self-report questionnaire that measures state anger, trait anger, expression and control of anger

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vidal, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Vidal R, Castells J, Richarte V, Palomar G, Garcia M, Nicolau R, Lazaro L, Casas M, Ramos-Quiroga JA. Group therapy for adolescents with attention-deficit/hyperactivity disorder: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2015 Apr;54(4):275-82. doi: 10.1016/j.jaac.2014.12.016. Epub 2015 Jan 26. PMID 25791144